CLINICAL TRIAL: NCT05516615
Title: The Predictive Value of the Heart Rate Response to Breathing Maneuvers for Inducible Myocardial Perfusion Deficits
Acronym: SCREEN-MORE
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Matthias Friedrich, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-6487
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: 1. Aged more than 35
  2. No known current or pre-existing problems that would affect the cardiovascular or respiratory system
  Interventions: Other: 4 minute breathing maneuver
- Patient population: 1. Aged more than 35
  2. Referral of subjects with known or suspected CAD for adenosine stress first-pass perfusion MRI based on the clinical judgement of their referring physician
  Interventions: Other: 4 minute breathing maneuver

INTERVENTIONS:
Other: 4 minute breathing maneuver — The 4-minute breathing maneuver comprised of 2 minutes of normal breathing and 1-min hyperventilation (rate of 30 breaths or more per minute) followed by a maximal breath-hold.

SUMMARY:
Breathing maneuvers, i.e. hyperventilation followed by breath-holding, have been shown to change coronary dynamics; hyperventilating narrows the coronary arteries, puts "stress" on the heart, and increases the heart rate, whereas breath-hold dilates the coronary arteries and decreases the heart rate," rest". Heart rate response to hyperventilation has been reported to have high diagnostic accuracy to rule out heart disease. The cardiac stress test, the modality of choice for the initial assessment of patients with suspected coronary artery disease(CAD), is routinely overprescribed by physicians, which exerts a financial burden on the healthcare system. Hence, developing an inexpensive, reliable, and available tool-HR response to breathing maneuvers- may avoid unnecessary referrals for cardiac stress tests by an effective differentiation of patients with CAD from healthy people. This study aims to assess the negative predictive value of the HR response to a 4-minute breathing maneuver for inducible myocardial ischemia, avoiding further stress testing as a gatekeeper.

DETAILED DESCRIPTION:
Patients with suspected CAD must have a clinical indication for cardiac stress test based on the clinical judgement of their referring physician and be referred to adenosine stress first-pass perfusion MRI located at the McGill University Health Centre (MUHC). Healthy participants must have no known history of cardiovascular or respiratory diseases. At the time of recruitment, eligible participants will perform the 4-minute breathing maneuver, comprised of 2 minutes of normal breathing and 1-min hyperventilation (rate of 30 breaths or more per minute) followed by a maximal breath-hold. A portable FDA-approved device will be used to record HR and respiration patterns during breathing maneuvers, which enables us to observe the beat-to-beat HR changes during each phase of the breathing maneuvers. On the same day, the participants' socio-demographics, medications, medical history and INTERHEART risk scores will be obtained. Afterwards, patients referred for a stress test will undergo adenosine stress first-pass perfusion MRI as prescribed by their referring physician to validate the findings of the breathing maneuver and detect CAD. Inside the MRI, the participants will also be asked to perform the same 4-min breathing maneuver during Oxygenation Sensitive-Cardiac Magnetic Resonance imaging (OS-CMR) protocol. This imaging technique provides a non-invasive assessment of myocardial oxygenation, relying on the paramagnetic features of deoxygenated hemoglobin as the intrinsic contrast agent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  1. Aged > 35
  2. No known current or pre-existing problems that would affect the cardiovascular or respiratory system

Patient population:

1. Aged > 35
2. Clinically indicated referral for adenosine stress first-pass perfusion MRI in subjects with known or suspected coronary artery disease

Exclusion Criteria:

Healthy Volunteers:

1. MR incompatible devices such as pacemakers, defibrillators, implanted material, or foreign bodies.
2. Consumption of caffeine (coffee, tea, cocoa, chocolate, "energy drink") during the 12 hours prior to the exam
3. Presence of cardiovascular disease.
4. Regular nicotine consumption during the last 6 months

Patient Population:

1. MR incompatible devices such as pacemakers, defibrillators, implanted material, or foreign bodies.
2. Vasoactive medication (e.g. nitrate, beta-blocker, calcium channel blocker) during the 12 hours prior to the exam.
3. Consumption of caffeine (coffee, tea, cocoa, chocolate, "energy drink") during the 12 hours prior to the exam
4. Acute Coronary Syndrome (ACS), or previous Coronary Artery Bypass Surgery
5. Previous myocardial infarction within one month
6. Clinically unstable condition
7. Significant or uncontrolled arrhythmia
8. Patients who are pregnant
9. Active myocarditis, constrictive pericarditis, any cardiomyopathy, cardiac or systemic amyloidosis
10. Left bundle branch block (LBBB)
11. Established valvular regurgitation or stenosis abnormality above moderate severity
12. Patients with a known history of heart failure (Ejection fraction<40%)

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with known or suspected Coronary Artery Disease (CAD) aged more than 35.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Assess the negative predictive value of the heart rate acceleration in response to 1-min hyperventilation | June 2020 - August 2021
  To rule out the presence of inducible myocardial perfusion deficit in patients with suspected coronary artery disease compared to healthy volunteers
  A ROC analysis will provide an optimal cut-point value for the level of heart rate acceleration in response to 1-min hyperventilation to identify its ability to rule out myocardial perfusion deficit
To assess the negative predictive value of the heart rate recovery in response to maximal voluntary breath-hold | June 2020 - August 2021
  To rule out the presence of inducible myocardial perfusion deficit in patients with suspected coronary artery disease compared to healthy volunteers
  A ROC analysis will provide an optimal cut-point value for the level of heart rate recovery in response to maximal voluntary breath-hold to identify its ability to rule out myocardial perfusion deficit

SECONDARY OUTCOMES:
To assess the negative predictive value of heart rate variability during 4-min breathing maneuver to rule out the presence of inducible myocardial perfusion deficit in patients with suspected coronary artery disease compared to healthy volunteers | June 2020 - August 2021
  ROC analysis will provide an optimal cut-point value for heart rate variability during 4-min breathing maneuver to identify its ability to rule out myocardial perfusion deficit
To assess the negative predictive value of the combination of INTERHEART risk score and HR response to breathing maneuver to rule out the presence of inducible myocardial perfusion deficit | June 2020 - August 2021
  ROC analysis will provide an optimal cut-point value for the combination of INTERHEART risk score and HR response to breathing maneuver to identify its ability to rule out myocardial perfusion deficit

OTHER OUTCOMES:
To compare the myocardial oxygenation changes in OS-CMR images between healthy volunteers and patients with suspected or known CAD | June 2020 - August 2021
  A student's t-test will compare the myocardial oxygenation changes between healthy volunteers and patients with suspected or known CAD
To assess the relationship between myocardial oxygenation changes in OS-CMR images with perfusion deficit in adenosine stress first-pass perfusion MRI | June 2020 - August 2021
  Pearson Correlation Coefficient will assess the correlation between myocardial oxygenation changes in OS-CMR with perfusion deficits in adenosine stress first-pass perfusion MRI

CONTACTS AND LOCATIONS:
Locations (1):
- The Research Institute of the McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No